CLINICAL TRIAL: NCT04429529
Title: Phase 1 First-in-Human, Time Lagged, Randomised, Placebo Controlled, Double Blind, Single Ascending Dose Study of TY027 in Healthy Adult Volunteers
Brief Title: Safety of TY027, a Treatment for COVID-19, in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tychan Pte Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCT-001
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-09

CONDITIONS: Coronavirus Disease-2019 (COVID-19)
Keywords: Coronavirus Disease-2019; COVID-19; SARS-CoV-2; Monoclonal Antibody; Infectious diseases; Phase 1 first in human study; Singapore
MeSH Terms: conditions — COVID-19; Communicable Diseases | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either treatment or placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- TY027 0.5 mg/kg (Experimental): Subject will be administered with 0.5 mg/kg of TY027 via IV infusion over a period of 30 minutes.
  Interventions: Biological: TY027
- Placebo 0.5 mg/kg (Placebo Comparator): Subject will be administered with 0.9% saline via IV infusion over a period of 30 minutes.
  Interventions: Other: 0.9% Saline
- TY027 5mg/kg (Experimental): Subject will be administered with 5 mg/kg of TY027 via IV infusion over a period of 30 minutes.
  Interventions: Biological: TY027
- Placebo 5 mg/kg (Placebo Comparator): Subject will be administered with 0.9% saline via IV infusion over a period of 30 minutes.
  Interventions: Other: 0.9% Saline
- TY027 10 mg/kg (Experimental): Subject will be administered with 10 mg/kg of TY027 via IV infusion over a period of 30 minutes.
  Interventions: Biological: TY027
- Placebo 10 mg/kg (Placebo Comparator): Subject will be administered with 0.9% saline via IV infusion over a period of 30 minutes.
  Interventions: Other: 0.9% Saline
- TY027 20 mg/kg (Experimental): Subject will be administered with 20 mg/kg of TY027 via IV infusion over a period of 30 minutes.
  Interventions: Biological: TY027
- Placebo 20 mg/kg (Placebo Comparator): Subject will be administered with 0.9% saline via IV infusion over a period of 30 minutes.
  Interventions: Other: 0.9% Saline
- TY027 30 mg/kg (Experimental): Subject will be administered with 30 mg/kg of TY027 via IV infusion over a period of 30 minutes.
  Interventions: Biological: TY027
- Placebo 30 mg/kg (Placebo Comparator): Subject will be administered with 0.9% saline via IV infusion over a period of 30 minutes.
  Interventions: Other: 0.9% Saline

INTERVENTIONS:
Biological: TY027 — TY027 Injection, (100 mg/5 mL/Vial), SARS-CoV-2 Monoclonal Antibody (mAb)
  Arms: TY027 0.5 mg/kg; TY027 10 mg/kg; TY027 20 mg/kg; TY027 30 mg/kg; TY027 5mg/kg
Other: 0.9% Saline — Placebo
  Arms: Placebo 0.5 mg/kg; Placebo 10 mg/kg; Placebo 20 mg/kg; Placebo 30 mg/kg; Placebo 5 mg/kg

SUMMARY:
The emergence and rapid spread of the coronavirus disease 2019 (COVID-19) since December 2019 across 188 countries globally has become a major public health crisis. COVID-19 was declared a pandemic by the World Health Organisation (WHO) on the 11th March 2020. To date, more than 14,000,000 cases and 600,000 deaths have been reported. COVID-19 is an acute respiratory disease caused by the novel SARS-CoV-2 virus from the Betacoronavirus genus, just like SARS-CoV and MERS-CoV. SARS-CoV-2 is primarily transmitted person-to-person through respiratory droplets or close contact. Fomite transmission has also been implicated as a transmission route. Common respiratory symptoms such as fever, sore throat, cough and shortness of breath, may appear 2 - 14 days after exposure. About 20% of infected cases progress to severe disease resulting in an estimated 2 - 5% mortality reported. With the unrelenting increase in cases being reported worldwide, there is thus an urgent need for therapeutics to be developed and used to disrupt the ongoing pandemic.

To date, there is no specific proven antiviral treatment for COVID-19. Supportive care is recommended for symptom relief and for severe cases, organ support is critical for optimal outcome. Numerous vaccine candidates against SARS-CoV-2 are under development and a couple have entered Phase 1 clinical trials. Remdesivir, a nucleotide analog, developed by Gilead Sciences as a treatment for Ebola virus disease is currently being repurposed and undergoing multiple clinical trials to evaluate safety and efficacy in COVID-19 patients. In a preliminary study, convalescent plasma containing neutralizing antibodies against SARS-CoV-2 has also been experimentally administered in critically ill COVID-19 patients with promising results. Donor plasma used was rich in virus specific IgG and IgM antibodies as determined by ELISA. Within days of convalescent plasma treatment, patients showed decrease in viral load (via qRT-PCR), as well as improved clinical status being observed. Tychan's TY027 will be the first biologics in the world, specifically targeting SARS-CoV-2, to enter human clinical trials. It is anticipated that a SARS-COV-2 specific monoclonal antibody therapeutic administered to acutely infected patients could reduce disease severity as well as prevent transmission by reducing viral load and viral shedding. It could also be used as prophylaxis against COVID-19 amongst high risk contacts.

DETAILED DESCRIPTION:
This is a Phase 1 First-in-Human, Time Lagged, Randomised, Placebo Controlled, Double Blind, Single Ascending Dose Study of TY027 in Healthy Adult Volunteers.

Safety, tolerability and PK of TY027 will be assessed. The dose escalation will include 32 healthy volunteers across five (5) dose cohorts:

* 0.5 mg/kg, N = 2 TY027 + 2 Placebos
* 5 mg/kg, N = 5 TY027 + 2 Placebos
* 10 mg/kg, N = 5 TY027 + 2 Placebos
* 20 mg/kg, N = 5 TY027 + 2 Placebos
* 30 mg/kg, N = 5 TY027 + 2 Placebos

Subjects will be required to be inpatient at the trial site for approximately 24 hours.

A minimum of 20-hour interval from the first two (2) subjects dosing (1 treatment and 1 placebo concurrently) must take place before the third subject can be dosed within the cohort. No such time interval will be required for dosing of subsequent subjects (fourth subject onwards) within the same dose cohort.

After 24 hours, subjects will be discharged from the trial site and to return for scheduled follow-up visits. Subjects will be followed for up to approximately Day 84 with serum samples taken at specified times as per outlines in Table 1.

Dose escalations will be guided by a safety review of clinical signs, adverse events (AEs), laboratory tests (excluding lipase) and immune gene expression data of the prior dose cohort (up to 72 hours post-dose). Subsequent post-trial monitoring through weekly telephone calls will continue from Day 85 onwards for another three (3) more months.

Decisions not to dose escalate past any proposed dose level due to safety findings will not constitute a protocol violation.

Safety summaries (up to Day 3 post-dose) will be generated for each dose cohort and delivered to the Dose Escalation Review Committee (DERC) for review.

Interim analysis will be performed after Day 14 post-dose for each dose cohort and delivered to the Data Safety Monitoring Board (DSMB) for review.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers, aged 21 to 50 years old, men or women
2. Subjects negative for human immunodeficiency virus (HIV antibody screen), Hepatitis B virus surface Antigen (HBsAg) and Hepatitis C virus (HCV antibody screen)
3. Subjects who are willing to comply with the requirements of the study protocol, attend scheduled visits and make themselves available for the duration of the study with access to a consistent means of telephone contact, which may be, but not limited to, at home or at work via landline or mobile
4. Subjects who give written informed consent approved by the Ethical Review Board governing the site
5. Satisfactory baseline medical assessment as assessed by physical examination and a stable health status. Normal laboratory values must be within normal range of the assessing site or show minor variations that are deemed not clinically significant as judged by the Investigator and acceptable for study entry. A stable health status is defined as the absence of a health event satisfying the definition of a serious adverse event
6. Accessible vein in the forearm for blood collection
7. Female subjects of childbearing potential may be enrolled in the study if they have negative urine pregnancy tests on the day of screening and day of admission
8. Female subjects of non-childbearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause. Post- menopause subjects must have had at least 12 months of natural (spontaneous) amenorrhea
9. Both male (if he has a partner of childbearing potential) and female subjects (of childbearing potential) must agree to use adequate and reliable contraceptive measures (e.g. spermicides, condoms, contraceptive pills, etc.) or practice abstinence throughout the duration of the study (up to 84 days post-dosing)

Exclusion Criteria:

1. Subject previously diagnosed with COVID-19 or had been issued with a quarantine order by the Ministry of Health
2. Presence of acute infection in the preceding 14 days, or presence of a temperature ≥ 38.0 ˚C (oral or tympanic temperature assessment), or acute symptoms of any severity on the scheduled date of admission
3. History of severe drug and / or food allergies and / or known allergies to the trial product or its components
4. Female subject who is pregnant or breast-feeding
5. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, neuropsychiatric, or immunosuppressive disorders
6. Evidence of clinically significant anaemia (HB < 10 g/dL) or any other significant active haematological disease, or having donated > 450 mL of blood within the past three (3) months
7. Participation or planned participation in a study involving the administration of an investigational compound within the past four (4) months or during this study period
8. Receipt of immunoglobulins and/or any blood products within nine (9) months of study enrolment or planned administration of any of these products during the study period
9. Administration of any licensed vaccine within 30 days before the first study vaccine dose.
10. History of any reaction to monoclonal antibodies
11. Any condition that, in the opinion of the Investigator, would complicate or compromise the study or well-being of the subject
12. Both male (if he has a partner of childbearing potential) and female subjects (of childbearing potential) who are unwilling to use adequate contraception or practice abstinence throughout the duration of the study (up to 84 days post-dosing)

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2020-11-19 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 84 Days
  To assess the safety and tolerability of an intravenous (IV) infusion of TY027 when administered to healthy adult volunteers. This will be assessed at various time points by clinical laboratory tests, vital signs and adverse events

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) - Pharmacokinetic Assessment | 84 Days
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the maximum concentration (Cmax) of TY027 in human serum.
Time to Maximum Concentration (Tmax) - Pharmacokinetic Assessment | 84 Days
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the time to maximum concentration (Tmax) of TY027 in human serum
Area Under the Curve Extrapolated to Infinity (AUC0-∞) - Pharmacokinetic Assessment | 84 Days
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the area under the curve extrapolated to infinity (AUC0-∞) of TY027.
AUC calculated from time of administration to the last measurable concentration (AUC0-last) - Pharmacokinetic Assessment | 84 Days
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the AUC calculated from time of administration to the last measurable concentration (AUC0-last) of TY027.
Half-Life (t1/2) - Pharmacokinetic Assessment | 84 Days
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the half-life (t1/2) of TY027 in human serum.
Volume of Distribution (Vd) - Pharmacokinetic Assessment | 84 Days
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the volume of distribution (Vd) of TY027 in human serum.
Clearance [CL] - Pharmacokinetic Assessment | 84 Days
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate clearance [CL] of TY027 in human serum.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Low, MBBS, Principal Investigator — SingHealth Investigational Medicine Unit
Locations (1):
- SingHealth Investigational Medicine Unit, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343